CLINICAL TRIAL: NCT03843970
Title: Hemodynamic Safety of Isobaric Levobupivacaine Versus Isobaric Bupivacaine for Subarachnoid Anesthesia in Patients Over 65 Years Undergoing Hip Surgery
Brief Title: Hemodynamic Safety of Levobupivacaine vs Bupivacaine in Patients Over 65 Years Undergoing Hip Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Clínico Universitario de Valencia (Other)
Responsible Party: Principal Investigator, ROSA HERRERA, MD, Principal Investigator, Hospital Clínico Universitario de Valencia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CoLeBu
Record Dates: First submitted 2018-05-28; First posted 2019-02-18 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Hip Fractures; Hemodynamic Stability
Keywords: Hip fracture, Subarachnoid block
MeSH Terms: conditions — Hip Fractures | interventions — dextran - saline drug combination; Elliott's solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Levobupivacaine Hydrochloride 0,5% (Experimental): The doses used of Levobupivacaine Hydrochloride 0.5% will be 6 mg and the dose of fentanyl 10 μg.
  Interventions: Drug: Levobupivacaine Hydrochloride 0.5%
- isobaric bupivacaine 0,5% (Active Comparator): The doses used of isobaric bupivacaine will be 6 mg and the dose of fentanyl 10 μg.
  Interventions: Drug: Isobaric bupivacaine 0.5%

INTERVENTIONS:
Drug: Levobupivacaine Hydrochloride 0.5% — The solution is called L solution, which contains a combination of 0.5% isobaric levobupivacaine with fentanyl. Injectable Solution.
  Other Names: L solution
  Arms: Levobupivacaine Hydrochloride 0,5%
Drug: Isobaric bupivacaine 0.5% — The solution is called B solution, which contains a combination of 0.5% isobaric bupivacaine with fentanyl. Injectable Solution.
  Other Names: B solution
  Arms: isobaric bupivacaine 0,5%

SUMMARY:
The altered hemodynamics, and therefore the arterial hypotension is the most prevalent adverse effect after subarachnoid anesthesia. The objective of the study was to determine the exact role of local anesthetic selection underlying spinal anesthesia-induced hypotension in the elderly patient. We conducted a descriptive, interventional pilot study to assess the hemodynamic impact of subarachnoid anesthesia with isobaric levobupivacaine versus isobaric bupivacaine for hip fracture surgery.

DETAILED DESCRIPTION:
1. Objective of the trial 1.1. Main objective: Compare the hemodynamic effects from invasive systolic diastolic and mean blood pressures (ISBP, IDBP and IMBP) mesured in mmHg, arterial partial pressure of oxygen (PaO2) and arterial partial pressure of carbon dioxide (PaCO2) measured in mmHg , arterial oxygen saturation (SatO2) measured in%, heart rate (HR / bpm) measured in beats per minute.

   Other variables of interest will be: cardiac index (CI) mesured in litres per minute per square metre (L/min/m2), peripheral vascular resistance (PVR) medured in dynes/seconds/cm-5, partial arterial pressure of oxygen (PaO2) and arterial partial pressure of carbon dioxide (PaCO2) measured in mmHg, pH (pH), arterial lactate (Lc) measured in mmol / L, arterial hemoglobin (Hb) measured in g/dl, partial oxygen saturation (SpO2%) measured in %.

   1.2. Secondary objectives: Assess potential adverse events during surgery and 48 hours of surgery. Adverse events include adverse cardiovascular and respiratory rate, events related to both surgical and anesthetic techniques and exitus.
2. End points 2.1. Primary end point(s): hemodynamic variables invasive systolic blood pressure (ISBP) measured in mmHg invasive diastolic blood pressure (ISBP), measured in mmHg invasive mean blood pressure (IMBP), measured in mmHg arterial partial pressure of oxygen (PaO2) arterial partial pressure of carbon dioxide (PaCO2), measured in mmHg arterial oxygen saturation (SatO2) measured in% heart rate (HR / bpm) measured in beats per minute cardiac index (CI) mesured in litres per minute per square metre (L/min/m2). peripheral vascular resistance (PVR) mesured in dynes/seconds/cm-5 partial arterial pressure of oxygen (PaO2) measured in mmHg arterial partial pressure of carbon dioxide (PaCO2) measured in mmHg pH (pH) arterial lactate (Lc) measured in mmol / L arterial hemoglobin (Hb) measured in g / dl partial oxygen saturation (SpO2%) measured in %.

2.1.1 Timepoint(s) of evaluation of this end point: entry into the operating room, after 30 minutes of anesthesia and at the end of anesthesia.

2.2. Secondary end point(s):

A. Intraoperative adverse events:

1. Cardiovascular and Respiratory: Venous air embolism (VAE), deep vein thrombosis (DVT), myocardial infarction (AMI), cerebrovascular accident (CVA), congestive heart failure (CHF), pneumonia (N), Exitus (Ex)
2. Other: Acute renal failure (ARF), vomiting (V)
3. Associated with the surgical technique: RBC transfusion (Th), plasma transfusion (TPL), nerve damage (ln), femur fracture (Fx f)
4. Associated with the anesthetic technique: paresthesia (pair), hematic puncture (ph), other.

B.Postoperative adverse events (at 48 hours)

1. Cardiovascular and Respiratory: Deep vein thrombosis (DVT), myocardial infarction (AMI), cerebrovascular accident (CVA), congestive heart failure (CHF), pneumonia (N), Exitus (Ex)
2. Other: Acute renal failure (ARF), UTI (Infu), vomiting (V).
3. Associated with the surgical technique: RBC transfusion (Th), plasma transfusion (TPL), neurologic deficit (defnq), surgical wound infection (Infhq).
4. Associated with the anesthetic technique: neurological deficit (defn), postdural puncture headache (PDPH), back pain (Lumb).

2.2.1. Timepoint(s) of evaluation of this end point: 48 hours of surgery

ELIGIBILITY:
Inclusion Criteria:

* Men and Women over 65 years
* Who meet the requirements in the pre-anesthetic to be treated with spinal anesthesia with levobupivacaine or bupivacaine, both with fentanyl,
* Fitness: from I to IV, according to the American Society of Anesthesiologists (ASA),
* Weight> 40 kg,
* Height> 140 cm,
* Body mass index (BMI) <50 kg/m2,
* Pathology cardiovascular, respiratory, renal and endocrine-metabolic,
* Provide written informed consent

Exclusion Criteria:

* Patients with uncontrolled hypertension (non-invasive systolic blood pressure> 180 mmHg and / or non-invasive diastolic blood pressure > 110mmHg),
* HR> 120 bpm,
* SpO2 <90% on arrival in the operating room and the contraindication to perform neuraxial anesthesia (patient refusal, infection at the site of puncture or lancing different, neuromuscular degenerative disease, hypovolemia, coagulopathy or anticoagulant therapy, morbid obesity, and extreme increase in intracranial pressure).

Ages: 65 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-06-14 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Compare hemodynamic effects from invasive systolic pressure, invasive diastolic pressure and mean blood pressure. | Intraoperative
  The measurement of invasive systolic pressure and invasive diastolic pressure and mean blood pressure mesured in mmHg.
Compare hemodynamic effects from heart rate. | Intraoperative
  The measurement of heart rate in beats per minute.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 48 hours of surgery
  Adverse events include adverse cardiovascular and respiratory rate, events related to both surgical and anesthetic techniques.

CONTACTS AND LOCATIONS:
Overall Officials: HERRERA ROSA, PhD, Principal Investigator — General University Hospital of Valencia
Locations (1):
- Hospital Clínico Universitario, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No